CLINICAL TRIAL: NCT01383148
Title: A Phase IIB/III Randomized, Double-blind, Placebo Controlled Study Comparing First Line Therapy With or Without TG4010 Immunotherapy Product in Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase IIB/III Of TG4010 Immunotherapy In Patients With Stage IV Non-Small Cell Lung Cancer
Acronym: TIME
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG4010.14/TIME; 8559 (Other: FDA)
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TG4010; Paclitaxel; Carboplatin; Pemetrexed; Cisplatin; Gemcitabine; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - TG4010 + first line therapy (Experimental): First-line therapy and maintenance therapy
  Interventions: Biological: TG4010
- Arm 2 : Placebo + first line therapy (Active Comparator): First-line therapy and maintenance therapy
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: TG4010 — TG4010 • TG4010 will be administered starting on Day 1 (D1) of Cycle 1 of chemotherapy and will be administered weekly for 6 weeks by subcutaneous (SC) injections and then once every 3 weeks until progression or discontinuation due to any reason.
  Chemotherapy (and bevacizumab if prescribed), will be given as 21-day cycles for a minimum of 4 cycles and up to 6 cycles.
  First line therapy:
  * Non-squamous carcinoma: pemetrexed + cisplatin or paclitaxel + carboplatin +/- bevacizumab
  * Squamous carcinoma: gemcitabine + cisplatin or paclitaxel + carboplatin
  Maintenance therapy:
  • Pemetrexed or erlotinib for eligible patients and according to labeling.
  Arms: Arm 1 - TG4010 + first line therapy
Drug: placebo — Placebo will be administered starting on D1 of Cycle 1 of chemotherapy and will be administered weekly for 6 weeks by SC injections and then once every 3 weeks until progression or discontinuation due to any reason.
  * First line therapy: as in Arm 1
  * Maintenance therapy: as in Arm 1
  Other Names: paclitaxel; carboplatin; pemetrexed; cisplatin; gemcitabine; bevacizumab (if prescribed); erlotinib
  Arms: Arm 2 : Placebo + first line therapy

SUMMARY:
This is a Phase IIb/III randomized, double-blind, placebo-controlled study to compare the efficacy and safety of first-line therapy combined with TG4010 or placebo in stage IV non-small cell lung cancer (NSCLC).

TG4010 is a suspension of recombinant Modified Vaccinia virus strain Ankara (MVA strain) carrying coding sequences for human MUC1 antigen and human interleukin-2 (IL2). TG4010 has been developed for use as an immunotherapy in cancer patients whose tumors express the MUC1 antigen.

TG4010 is intended to induce a MUC1-specific cellular immune response and to produce a non-specific activation of several components of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma, undifferentiated carcinoma or other)
* Stage IV cancer according to TNM classification (7th edition - UICC, December 2009; includes tumor with malignant pleural or pericardial effusion
* Tumor biopsy specimen with ≥ 50% of MUC1 expressing tumor cells determined by Immunohistochemistry (IHC) staining on fixed pathological material. Biopsy may come either from the primary tumor or from a metastasis. Cytological material is not accepted for this analysis
* Patient's naïve to first-line therapy for the advanced stage of the disease. Previous neoadjuvant or adjuvant therapy is allowed for patients who successfully underwent complete radical surgery and if last treatment was administered more than 12 months prior to the start of the study treatment, i.e., D1 of Cycle 1.
* At least one measurable lesion by CT scan or MRI based on RECIST version 1.1
* PS 0 or 1 on the ECOG scale
* Adequate hematological, hepatic, and renal function:

  * Hemoglobin ≥ 10.0 g/dL
  * White Blood Cells (WBC) ≥ 3.0x10E9/L including

    * Neutrophils ≥ 1.5x109/L
    * Total lymphocytes count ≥ 0.5x10E9/L
  * Platelets count ≥ 100x10E9/L
  * Serum alkaline phosphatase ≤ 3x ULN (upper limit of normal)in the absence of liver or bone metastases or ≤5 ULN(in patients with documented bone or liver metastases)
  * Serum transaminases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) ≤ 2.5 x ULN in the absence of liver metastases or =< 5 ULN in case of liver metastases)
  * Total bilirubin ≤1.5 x ULN
  * Glomerular Filtration Rate ≥ 60 mL/min (according to Modification of the Diet in Renal Disease (MDRD) formula or cockroft & Gault formula)
  * Serum albumin ≥ 30 g/L
  * Effective contraception during the study period and for 3 months after the last study treatment administration (male and female patient)

Exclusion Criteria:

* Patients having Central Nervous System (CNS) metastases. Patients who have had brain metastases surgically removed or irradiated with no residual disease confirmed by imaging are allowed
* Documented EGFR activating mutations (if already tested)
* Prior history of other malignancy except:

  * Basal cell carcinoma of the skin
  * Cervical intra epithelial neoplasia
  * Other cancer curatively treated with no evidence of disease for at least 5 years
* Patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (e.g., cyclosporine) for a period of at least 4 weeks and whose treatment was not stopped 1 week prior to the start of the study treatment (i.e., D1 of Cycle 1)
* Positive serology for Human Immunodeficiency Virus (HIV) or Hepatitis C Virus (HCV); presence in the serum of the antigens HBs
* Patient with any underlying medical condition that the treating physician considers might be aggravated by treatment or which is not controlled (e.g., elevated troponin or creatinine, uncontrolled diabetes)
* Patient with major surgery or radiotherapy within 4 weeks prior to the start of the study treatment (i.e., D1 of Cycle 1). Prior surgery or radiation therapy aimed at local palliation or attempted local disease control is permitted
* Patient with an organ allograft
* Known allergy to eggs, gentamicin or platinum-containing compounds
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatment (i.e., D1 of Cycle 1)
* Patient unable or unwilling to comply with the protocol requirements
* Pregnancy or lactation
* Bevacizumab will be allowed for patients with non-squamous carcinoma. Prescribing information must be followed and precautions have to be taken into consideration (e.g., patients having presented a serious hemorrhage or recent hemoptysis should not receive bevacizumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-04; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Phase 2: Progression-free Survival (PFS) | Approximately 15 months
  PFS is measured from date of randomization to radiographically documented progression according to RECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Phase 3: Overall Survival (OS) | Approximately 27 months
  OS is measured from date of randomization to date of death from any cause.

SECONDARY OUTCOMES:
Phase 2 : Overall Survival (OS) | Approximately 15 months
Phase 2 : Overall Response Rate (ORR) | Approximately 15 months
Phase 3: Progression-free Survival (PFS) | Approximately 27 months
Phase 3 : Overall Response Rate (ORR) | Approximately 27 months
Phase 2 : Duration of response | Approximately 15 months
Phase 2: Safety | Approximately 15 months
Phase 3: Duration of response | Approximately 27 months
Phase 3: Safety | Approximately 27 months

CONTACTS AND LOCATIONS:
Overall Officials: QUOIX Elisabeth, Prof, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (72):
- United States (12):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Cambridge, Maryland
  - Oncology/Hematology P.C., Rockville, Maryland
  - Washington University, St Louis, Missouri
  - Highlands Oncology Group, Fayetteville, North Carolina
  - Signal Point Clinical Research Center, Middletown, Ohio
  - ProMedica Health System Inc, Toledo, Ohio
  - Abington Hematology Oncology Associates Inc, Willow Grove, Pennsylvania
  - Texas Oncology, P.A. - Abilene (South), Abilene, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Clinique Nôtre-Dame de Grâce, Gosselies
  - Centre Hospitalier de l'Ardenne, Libramont
  - C. H. U. Sart-Tilman, Liège
- France (16):
  - CHU, Service de Pneumologie, Besançon
  - Centre François Baclesse, Caen
  - CHU de Clermont-Ferrand, Hopital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Pasteur - Service de médecine F- Pavillon 43, Colmar
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHRU de Lille Hopital Calmette, Lille
  - Clinique François Chénieux, Limoges
  - Institut Paoli-Calmettes, Service d'oncologie médicale, Marseille
  - CH Mulhouse Hopital Emile Muller Moenchsberg, Mulhouse
  - Hopital Saint Joseph, Paris
  - Hôpital Pontchaillou, Rennes
  - CHU de Saint-Etienne, Hôpital Nord, Saint-Etienne
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Médical Alfred Leune, Sainte-Feyre
  - Nouvel Hôpital Civil, Strasbourg
  - Centre Hospitalier Intercommunal de la Haute Saone, Vesoul
- Germany (2):
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Mannheim, Mannheim
- Hungary (12):
  - Orszagos Onkologiai Intezet, Budapest
  - Semmelweis Egyetem AOK, Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Kenezy Korhaz-Rendelointezet Eu Szolgaltato Nonprofit Kft, Debrecen
  - Petz Aladár Megyei Oktató kórház, Győr
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Gyula
  - Matrai Gyogyintezet, Mátraháza
  - Tolna Megyei Onkormanyzat Balassa Janos Korhaza, Szekszárd
  - Fejér Megyei Szent György Kórház, Székesfehérvár
  - Komarom-Esztergom Megyei Onkorm. Szent Borbala Korhaza, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Korhaz, Zalaegerszeg
- Israel (7):
  - Assaf Harofeh Medical Center, Beer Yaacov
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Sapir Medical Center Meir Hospital, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera di Perugia Ospedale S.Maria della Miseri, Perugia
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Poland (5):
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - SP Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - ICO Girona - Hospital Dr Josep Trueta, Girona
  - Hospital Gregorio Marañon, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid
  - Hospital General Carlos Haya, Málaga
  - Corporació Sanitària Parc Taulí, Sabadell
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Hospital NHS Trust, Cardiff
  - Plymouth Oncology Centre, Plymouth
  - Southampton University Hospitals NHS Trust, Southampton

REFERENCES:
- [Derived] Tosch C, Bastien B, Barraud L, Grellier B, Nourtier V, Gantzer M, Limacher JM, Quemeneur E, Bendjama K, Preville X. Viral based vaccine TG4010 induces broadening of specific immune response and improves outcome in advanced NSCLC. J Immunother Cancer. 2017 Sep 19;5(1):70. doi: 10.1186/s40425-017-0274-x. PMID 28923084
- [Derived] Quoix E, Lena H, Losonczy G, Forget F, Chouaid C, Papai Z, Gervais R, Ottensmeier C, Szczesna A, Kazarnowicz A, Beck JT, Westeel V, Felip E, Debieuvre D, Madroszyk A, Adam J, Lacoste G, Tavernaro A, Bastien B, Halluard C, Palanche T, Limacher JM. TG4010 immunotherapy and first-line chemotherapy for advanced non-small-cell lung cancer (TIME): results from the phase 2b part of a randomised, double-blind, placebo-controlled, phase 2b/3 trial. Lancet Oncol. 2016 Feb;17(2):212-223. doi: 10.1016/S1470-2045(15)00483-0. Epub 2015 Dec 23. PMID 26727163
- See also: NSCLC — http://www.ncbi.nlm.nih.gov/pubmed?term=nsclc
- See also: Therapeutic vaccination with TG4010 and first-line chemotherapy in advanced non-small-cell lung cancer: a controlled phase 2B trial., Lancet Oncol. 2011 Nov;12(12):1125-33. Epub 2011 Oct 21. — http://www.ncbi.nlm.nih.gov/pubmed/22019520